CLINICAL TRIAL: NCT02153736
Title: Initial Efficacy Study of Supporting Play, Exploration, & Early Development Intervention (SPEEDI) - Phase 1 Clinical Trial
Brief Title: Initial Efficacy Study of Supporting Play, Exploration, & Early Development Intervention
Acronym: SPEEDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Foundation for Physical Therapy, Inc. (Industry); Children's Hospital Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM20001308
Record Dates: First submitted 2014-05-27; First posted 2014-06-03 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Infant, Premature, Diseases; Brain White Matter Disease Periventricular
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Group (No Intervention): This group of subjects will receive usual care provided in the medial system and community.
- SPEEDI Intervention (Experimental): This group will receive and parent and physical therapy provided intervention to increase the infants opportunities for play which will enhance development.
  Interventions: Behavioral: SPEEDI Intervention

INTERVENTIONS:
Behavioral: SPEEDI Intervention — Behavioral intervention provided through a collaboration between the mother of enrolled subjects and a physical therapist. Intervention starts in the Neonatal Intensive Care Unit and continues after discharge. SPEEDI includes both parent education and developmental activities.
  Arms: SPEEDI Intervention

SUMMARY:
The primary aims of this randomized controlled trial are to evaluate efficacy potential of SPEEDI at enhancing reaching and play based problem solving compared to infants receiving usual care.

DETAILED DESCRIPTION:
The primary aims of this randomized controlled trial are to evaluate efficacy potential of SPEEDI at enhancing reaching and play based problem solving compared to infants receiving usual care. The secondary aim is to assess the efficacy potential of SPEEDI to impact motor and cognitive development as assessed using commonly used clinical outcome measures. The exploratory aims are to assess the impact of SPEEDI on parent child interactions and feeding skills. The findings will provide crucial initial efficacy estimates to be used in a larger definitive clinical trial of SPEEDI.

ELIGIBILITY:
Inclusion Criteria:

* born extremely preterm (˂29 weeks of gestation) OR 10 born preterm and diagnosed with a neonatal brain injury including intraventricular hemorrhage grade 3 or 4, periventricular white matter injury, or hydrocephalus requiring a shunt.
* Medically stable by 40 weeks of gestation, including being off ventilator support
* Live within 50 minutes of the hospital.
* English Speaking mother
* Mother willing and able to participate in the study with the infant subject

Exclusion Criteria:

* Genetic syndromes or musculoskeletal deformities

Max Age: 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey C Dusing, PhD PT, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Given the small sample from a specific time range the data will not be shared due to difficulty de-identifying with demographics of individual infants attached.

REFERENCES:
- [Derived] Dusing SC, Tripathi T, Marcinowski EC, Thacker LR, Brown LF, Hendricks-Munoz KD. Supporting play exploration and early developmental intervention versus usual care to enhance development outcomes during the transition from the neonatal intensive care unit to home: a pilot randomized controlled trial. BMC Pediatr. 2018 Feb 9;18(1):46. doi: 10.1186/s12887-018-1011-4. PMID 29426320

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care Group | SPEEDI Intervention
Started | 7 | 7
Completed | 5 | 5
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Medical status change made ineligible | 1 | 0
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Group | SPEEDI Intervention | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Median (Inter-Quartile Range); unit: Weeks of post menstrual age] | 35 [35 to 39] | 39 [36 to 40] | 38 [35 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 1 | 1 | 2
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14
Gestational age [Median (Inter-Quartile Range); unit: weeks of gestation] | 26 [25 to 28] | 25 [24 to 27] | 25.5 [25 to 27]
Brain Injury (GIII/IV intraventricular hemorrhage , Periventricular leukomalacia, Hypoxic Ischemic E [Count of Participants; unit: Participants] — Clinical cranial ultrasound in the neonatal period was used to document the presence of any reported intraventricular hemorrhage or periventricular leukomalacia as all included infants meet the clinical guidelines for having a cranial ultrasound in the neonatal intensive care unit. Radiology reports including a finding of Grade III/IV (severe) intraventricular hemorrhage, periventricular leukomalacia, or Diffuse brain injury were used to stratify infants into a severe brain injury group
  Participants | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Reaching (Toy Contact Duration)
Description: Duration the infant is in contact with the target is used to quantify changes in reaching.
Time Frame: 1 month post intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Usual Care Group | SPEEDI Intervention
Number analyzed (Participants) | 5 | 5
Seconds | 20.2 (21.45) | 28.02 (16.30)

2. Primary Outcome: Early Problem Solving Indicator (EPSI)
Description: Problem-solving behaviors were assessed using the Early Problem Solving Indicator (EPSI). The EPSI is the cognitive subtest of the Individual Growth and Development Indicators designed to measure infant and toddler play-based problem-solving through 36 months of age. It defines problem-solving as consisting of visual exploration, object manipulation and memory. The infant was video-recorded interacting with 3 standard toys: pop-up animals toy, 6 seriated, plastic cups, and a gum ball machine with 5 balls. Infants were given each toy for 2 minutes. The frequency of 4 mutually exclusive behaviors (look, explore, function, solution) were coded using definitions from the EPSI protocol. time. The total number of problem solving behaviors was calculated as a sum of look, explore, function, and solution for each infant at each visit and reported as the total EPSI frequency with a higher frequency reflecting more problem solving behaviors.
Time Frame: End of intervention, 1 and 3 months post intervention
Population: Same as primary population with the 2 infants lost to follow up not included.
Measure: Mean (Standard Deviation); unit: # of Problem Solving Behaviors in 6 min
Arm/Group | Usual Care Group | SPEEDI Intervention
Number analyzed (Participants) | 5 | 5
# of Problem Solving Behaviors in 6 min
  End of intervention | 58.00 (39.59) | 103.2 (28.89)
  1 months post intervention | 95.2 (52.95) | 131.80 (61.44)
  3 months post intervention | 146 (86.17) | 212 (54.98)

3. Secondary Outcome: Early Feeding Skill Assessment (FES)
Description: The Early Feeding Skills (EFS) was used to assess the infant's oral feeding skills during the video recorded feeding described above. The EFS is a 26-item observational tool that can be used from the start of oral feeding through the maturation of feeding skills. Each item can score 1-3 with one representing the least skill or high frequency of problem (an area of clinical concern), and three representing mature skill or absence of problem (area of strength). Subscales included were ability to maintain engagement in feeding, ability to organize oral-motor functioning, ability to coordinate swallowing, and ability to maintain physiological stability. The sum of all the items in a subscale divided by the number of items in the subscale gives the subscale score of 1-3. The sum of all subscales was used to create an EFS total score which could range from 2 to 12 with a higher score reflecting a better feeding performance.
Time Frame: Baseline, End phase 1, End of intervention, 1 and 3 months post intervention
Population: Some infants were not able to orally feed in which case this measure was not included. In addition, some visits were missing feeding assessments for missing data. Thus the sample included varied some between visits.
Measure: Mean (Standard Deviation); unit: EFS Total score
Arm/Group | Usual Care Group | SPEEDI Intervention
Number analyzed (Participants) | 6 | 6
EFS Total score
  Baseline: number analyzed (Participants) | 4 | 6
  Baseline | 8.32 (.48) | 8.61 (1.44)
  End phase 1: number analyzed (Participants) | 6 | 5
  End phase 1 | 8.27 (1.27) | 8.82 (1.58)
  End of intervention Phase 2: number analyzed (Participants) | 3 | 5
  End of intervention Phase 2 | 8.00 (0.44) | 9.65 (1.17)
  1 month post intervention: number analyzed (Participants) | 4 | 4
  1 month post intervention | 10.10 (1.36) | 9.91 (1.12)
  3 months post intervention: number analyzed (Participants) | 3 | 3
  3 months post intervention | 10.00 (1.42) | 10.40 (1.57)

4. Secondary Outcome: Parent Child Early Relational Assessment (PCERA)
Description: The Parent-Child Early Relational Assessment (PCERA; Clark, 2010; Clark, 1999) was designed to assess mother-infant interaction. In this study PCERA was scored from a video of the feeding interaction. The PCERA is a 65-item observational rating scale (29 parental, 27 infant, and 8 dyadic), designed to assess the amount, duration, and intensity of interaction. Each item was rated on a 3-point ordinal scale with 1-2 indicating an area of concern, 3 indicating an area for some concern and 4- 5 indicating an area of strength. Eight subscales constructed from items of the PCERA have been theoretically derived and confirmed by factor analysis (Clark, 1999; Clark et al., 1997). For ease of analysis this scale was transformed to a -1 to +1 range. Scores were recorded as 1 or 2 = -1, 3= 0, 4 or 5 = 1. The total PCERA score is the mean of all the subscale mean scores and ranged -1 (highest risk of atypical interactions) to +1 (most positive interactions).
Time Frame: Baseline, End phase 1, End of intervention, 1 month post intervention
Population: The sample varied some between visits do to a lack of video taping the parent child interaction on a few occasions because the parent who consented to the study was not present at the time of the visit and the visit could not be rescheduled. The 3 month post intervention visit was dropped.
Measure: Mean (Standard Deviation); unit: Mean Score on PCERA
Arm/Group | Usual Care Group | SPEEDI Intervention
Number analyzed (Participants) | 6 | 6
Mean Score on PCERA
  Baseline: number analyzed (Participants) | 6 | 4
  Baseline | 0.27 (0.17) | 0.13 (0.29)
  End phase 1: number analyzed (Participants) | 5 | 5
  End phase 1 | 0.20 (0.30) | 0.38 (0.33)
  End of intervention Phase 2: number analyzed (Participants) | 3 | 5
  End of intervention Phase 2 | 0.34 (0.24) | 0.25 (0.23)
  1 months post intervention: number analyzed (Participants) | 2 | 4
  1 months post intervention | 0.50 (0.51) | 0.26 (0.25)

5. Secondary Outcome: Bayley Scales of Infant and Toddler Development (Bayley).
Description: The Bayley-III is a norm references standardized developmental assessment of Motor, Cognitive, and Language skills. Composite scores for each domain have a mean of 100 and a standard deviation of 15. A score of 85-115 is considered average. Higher composite scores represent higher or better performance on that subtest. The Bayley was administered at the final follow-up visit and 3 months after the intervention ended.
Time Frame: 3 month post intervention
Population: At 3 months post intervention the sample was consistent with that described in the study sample post lose to followup.
Measure: Mean (Standard Deviation); unit: Mean Composite Score on Bayley
Arm/Group | Usual Care Group | SPEEDI Intervention
Number analyzed (Participants) | 5 | 5
Mean Composite Score on Bayley
  Motor 3 months post intervention | 79.6 (20.8) | 98.6 (11.4)
  Cognitive 3 months post intervention | 80.0 (13.5) | 91.0 (8.9)
  Language 3 months post intervention | 89.0 (19.6) | 98.2 (9.6)

6. Secondary Outcome: Test of Infant Motor Performance (TIMP)
Description: The TIMP is a standardized and norm references test of motor control and posture in infants 4 months of age and younger which is commonly used with infants starting at 34 weeks of post-menstrual age. Change in raw score from baseline to end of the intervention is reported. The TIMP raw score ranges from 0 to 142. A higher score represented greater performance in motor control and posture.
Time Frame: Baseline to End of intervention
Population: Full Sample after infants lost to follow up who are not included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Raw Score on the TIMP
Arm/Group | Usual Care Group | SPEEDI Intervention
Number analyzed (Participants) | 5 | 5
Raw Score on the TIMP
  Baseline | 54 [37 to 60] | 61 [56 to 63]
  End of Intervention | 82 [72 to 95] | 99 [97 to 118]

ADVERSE EVENTS:
Arm/Group | Usual Care Group | SPEEDI Intervention
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
Sample smaller than anticipated Fewer infant with brain injury than anticipated ceiling effect notes with reaching measures longer term outcomes only possible from clinical records

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No